CLINICAL TRIAL: NCT00268879
Title: A Phase III Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of Renzapride in Women With Constipation-Predominant Irritable Bowel Syndrome (c-IBS)
Brief Title: Investigation of the Safety and Efficacy of Renzapride in Constipation Predominant Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alizyme (Industry)
Responsible Party: Research and Development Director, Alizyme
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATL1251/038/CL
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Constipation-predominant irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — renzapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Two capsules are taken by mouth each morning and each evening from the day of the randomization visit until the scheduled visit at the end of Week 12.
  Interventions: Drug: Renzapride
- 2 (Experimental): Renzapride 4 mg QD. Two capsules are taken by mouth each morning and each evening from the day of the randomization visit until the scheduled visit at the end of Week 12.
  Interventions: Drug: Renzapride
- 3 (Experimental): Renzapride 2 mg BID: Two capsules are taken by mouth each morning and each evening from the day of the randomization visit until the scheduled visit at the end of Week 12.
  Interventions: Drug: Renzapride

INTERVENTIONS:
Drug: Renzapride — Placebo Renzapride 4 mg QD Renzapride 2 mg BID
  Other Names: ATL-1251; BRL-24924

SUMMARY:
The purpose of the study is to investigate whether renzapride will help alleviate the symptoms associated with constipation predominant irritable bowel syndrome in female patients.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic gastrointestinal disorder characterized by recurrent symptoms of abdominal pain/discomfort accompanied by disturbed bowel function.

In this study female patients with constipation predominant IBS will receive one of two dosing regimens of renzapride or placebo for 12 weeks. Patients will record the severity of their symptoms throughout the study. The results will be analysed to see if those patients who received renzapride had greater relief of their symptoms than did the patients who received placebo.

ELIGIBILITY:
Inclusion Criteria:

* Females with constipation predominant IBS as defined by the Rome II criteria
* Colonoscopy or sigmoidoscopy in previous 5 years showed no significant disease

Exclusion Criteria:

* Patients who have diarrhoea predominant or alternating symptom IBS
* Other gastrointestinal diseases that affect bowel transit

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1821 (Actual)
Dates: Start 2005-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Number of months a patient is a Responder for overall relief of IBS symptoms | 12 weeks

SECONDARY OUTCOMES:
Number of months a patient is a Responder for relief of abdominal pain/discomfort, bowel problems, and bloating/abdominal distention | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lembo, Principal Investigator — Beth Israel Deaconess Medical Centre, Boston
Locations (1):
- Alizyme, Cambridge, United Kingdom